CLINICAL TRIAL: NCT00210041
Title: Phase 2 Study for Treatment of Penis Epidermoid Carcinoma Loco-regionally Advanced or Metastatic by Association Gemcitabine-Cisplatin
Brief Title: Phase 2 Study of Association Gemcitabine-Cisplatin to Treat Penis Epidermoid Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03 GENH 06; 02 GENM 02
Record Dates: First submitted 2005-09-02; First posted 2005-09-21 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Genital Neoplasms, Male
Keywords: Genital Neoplasms, Male
MeSH Terms: conditions — Genital Neoplasms, Male | interventions — Gemcitabine; Cisplatin

INTERVENTIONS:
Drug: Gemcitabine — Gemzar IV infusion 30 minutes Day 1/ Day 15 1250 mg/m²/j
Drug: Cisplatin — Cisplatin 50 mg/m²/day 1 h IV infusion at Day 1 / Day 15

SUMMARY:
The purpose of this study is to determine whether association Gemcitabine-Cisplatin is effective in the treatment of penis epidermoid carcinoma loco-regionally advanced or metastatic.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* OMS ≤ 2
* Penis epidermoid carcinoma histologically proved. Tumor with ganglionic loco-regional injury inextirpable and/or metastatic (M1, all T , all N), at initial diagnostic or at relapse after first treatment with curative aim (surgery and / or radiotherapy)
* Disease measurable with RECIST criteria
* Absence of all former chemotherapy during 5 years between inclusion.
* If former radiotherapy, necessity to have appreciated targets outside the irradiation fields. If former radiotherapy, it must have been done more than 4 weeks before inclusion in the study.
* Biologicals values required : polynuclear neutrophils ≥ 1500/mm3, blood-platelets ≥ 100000/mm3, Hb ≥ 10 g/dl, Transaminases < 3N, TP ≥ 70%, total bilirubin < 1,5 N, creatinine in the blood ≤ 110 micromoles/l.
* Normal clearance of creatinine, according to Cockroft and Gault's formulae.
* Calcemia : normal or anomaly without clinical meaning.
* Well-informed written consent, signed by the patient.

Exclusion Criteria:

* Uncontrolled cerebral known metastasis
* All former chemotherapy administration during 5 years between inclusion
* Other cancer (except baso-cellular cancer of skin correctly treated, or cancerous disease considered with good prognosis and on remission until 5 years at least)
* Uncontrolled cardiac insufficiency or all other severe and uncontrolled pathology.
* Peripheric neuropathy ≥ grade 2 OMS
* Anormal audiogram
* Patient difficult to follow for geographical, psychological or family reasons.
* Persons protected by law.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-02; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To evaluate objective response rate | until desease progression

SECONDARY OUTCOMES:
To evaluate tolerance of the association, | during all participation of the subject
time to progression, | untill progression
global survival | untill death

CONTACTS AND LOCATIONS:
Overall Officials: Christine Chevreau, Doctor, Principal Investigator — Institut Claudius Regaud
Locations (11):
- France (11):
  - Centre Paul Papin, Angers
  - Institut Bergonie, Bordeaux
  - Centre François Baclesse, Caen
  - CHU Grenoble, Grenoble
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmette, Marseille
  - Institut Val d'aurelle, Montpellier
  - Institut Curie, Paris
  - Centre Eugène Marquis, Rennes
  - Centre Médico-Chirurgical Foch, Suresnes
  - Institut Claudius Regaud, Toulouse